CLINICAL TRIAL: NCT02195687
Title: BOTOX® in the Treatment of Crow's Feet Lines in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622-113
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Lateral Canthal Lines; Crow's Feet Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin type A (Experimental): 24U botulinum toxin Type A (BOTOX®) total dose injected into bilateral Crow's Feet Line areas on Day 1.
  Interventions: Biological: botulinum toxin Type A
- placebo (Placebo Comparator): Placebo (Normal Saline) injected into bilateral Crow's Feet Line areas on Day 1.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A (BOTOX®) injected into bilateral crow's feet line areas.
  Other Names: BOTOX®
  Arms: botulinum toxin type A
Drug: Normal Saline — Normal Saline (placebo) injected into bilateral Crow's Feet Line areas.
  Arms: placebo

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® (botulinum toxin Type A) compared with placebo in patients with moderate to severe crow's feet lines (lateral canthal lines).

ELIGIBILITY:
Inclusion Criteria:

-Moderate to severe Crow's Feet Lines.

Exclusion Criteria:

* Current or previous treatment with botulinum toxin of any serotype for any condition within the last year
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis
* Facial laser or light treatment, microdermabrasion or chemical peels within 3 months
* Radio frequency laser treatments, phototherapy, blepharoplasty, brow-lift or related procedure, permanent make-up, oral retinoid therapy or treatment with non-permanent soft tissue fillers within 1 year
* Any medium-depth or deep facial peels within 5 years
* Periorbital surgery, face-lift, mid facial or periorbital treatment with permanent soft tissue fillers, synthetic implants or autologous fat transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Beijing, China

REFERENCES:
- [Derived] Wu Y, Li C, Garcia J, Baradaran S. Patient-reported Outcomes in Chinese Subjects Treated with OnabotulinumtoxinA for Crow's Feet Lines. J Clin Aesthet Dermatol. 2021 Oct;14(10):27-31. PMID 34976286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant flow reflects the Safety Population, which includes all randomized subjects who received at least 1 study drug injection.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Placebo
Started | 316 | 101
Completed | 311 | 99
Not Completed | 5 | 2
Not completed — Personal Reasons | 1 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo | Total
Number analyzed (Participants) | 316 | 101 | 417
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (9.64) | 46.6 (9.39) | 46.4 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 87 | 360
  Male | 43 | 14 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving None or Mild on the Investigator's Assessment of the Severity of Crow's Feet Lines (CFL) at Maximum Smile Using the Facial Wrinkle Scale-Asian (FWS-A)
Description: The Investigator assessed the severity of the subject's CFLs at maximum smile using the 4-point FWS-A where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of subjects with a score of none or mild at Day 30 is reported.
Time Frame: Day 30
Population: Modified Intent-to-Treat: all randomized subjects who received at least 1 injection of study drug
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 316 | 101
Percentage of Subjects | 63.9 | 5.0

2. Secondary Outcome: Percentage of Subjects With a ≥ 1-grade Improvement on the Investigator's Assessment of CFL Severity at Rest Using the 4-point FWS-A
Description: The Investigator assessed the severity of the subject's CFLs at rest using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe among subjects rated as at least mild at baseline by the Investigator. The percentages of subjects with at least a 1-grade improvement are noted.
Time Frame: Day 30
Population: Modified Intent-to-Treat: all randomized subjects who received at least 1 injection of study drug
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 316 | 101
Percentage of Subjects | 60.1 | 5.4

3. Secondary Outcome: Percentage of Subjects With a ≥ 1-grade Improvement on the Investigator's Assessment of CFL Severity at Maximum Smile on the 4-point FWS-A
Description: The Investigator assessed the severity of the subject's CFLs at maximum smile using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe. The percentages of subjects with at least a 1-grade improvement are noted.
Time Frame: Day 30
Population: Modified Intent-to-Treat: all randomized subjects who received at least 1 injection of study drug
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 316 | 101
Percentage of Subjects | 85.1 | 12.9

4. Secondary Outcome: Percentage of Subjects Reporting Their Global Change in Appearance as Very Much Improved or Much Improved Using the 7-point Subject's Global Assessment of Change in CFL (SGA-CFL)
Description: Subjects assessed their global change in appearance using the 7-point SGA-CFL scale where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The percentage of subjects reporting very much improved or much improved are noted.
Time Frame: Day 30
Population: Modified Intent-to-Treat: all randomized subjects who received at least 1 injection of study drug
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 316 | 101
Percentage of Subjects | 54.4 | 3.0

5. Secondary Outcome: Percentage of Subjects Assessing Their Age-related Facial Appearance as Looking Younger on the Self-Perception of Age (SPA) Questionnaire
Description: Subjects assessed their age-related appearance according to the following on the SPA questionnaire: look my current age, look younger, and look older when compared to their baseline assessment. The percentages of subjects who reported looking younger amongst subjects who rated themselves as looking their current age or older at baseline are noted.
Time Frame: Baseline, Day 30
Population: Modified Intent-to-Treat: all randomized subjects who received at least 1 injection of study drug and rated themselves as looking their current age or older at baseline
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 297 | 95
Percentage of Subjects | 53.9 | 14.7

6. Secondary Outcome: Percentage of Subjects Achieving None or Mild on the Subject's Assessment of the Severity of Crow's Feet Lines (CFL) at Maximum Smile Using the Facial Wrinkle Scale-Asian (FWS-A)
Description: The subject assessed the severity of their CFLs at maximum smile using the 4-point FWS-A where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of subjects with a score of none or mild at Day 30 is reported.
Time Frame: Day 30
Population: Modified Intent-to-Treat: all randomized subjects who received at least 1 injection of study drug
Measure: Number; unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 316 | 101
Percentage of Subjects | 60.8 | 5.9

ADVERSE EVENTS:
Description: The Safety Population included all randomized subjects who received at least 1 study drug injection. The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Botulinum Toxin Type A | Placebo
Serious Adverse Events (participants affected / at risk) | 0/316 | 0/101
Other Adverse Events (participants affected / at risk) | 0/316 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.